CLINICAL TRIAL: NCT00002852
Title: A PHASE III STUDY OF ADJUVANT CHEMOTHERAPY AFTER RESECTION FOR PATIENTS WITH T2N0 STAGE I NON-SMALL CELL CARCINOMA OF THE LUNG
Brief Title: Surgery With or Without Chemotherapy in Treating Patients With Stage I Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02967; CALGB-9633; CDR0000065095; CLB-C9633; U10CA031946 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Bronchoalveolar Cell Lung Cancer; Large Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Taxes; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (surgery, observation) (Active Comparator): Patients receive no further therapy.
  Interventions: Procedure: therapeutic conventional surgery
- Arm II (surgery, chemotherapy) (Experimental): Patients receive adjuvant therapy comprising paclitaxel IV over 3 hours followed by carboplatin IV over 1-2 hours on day 1. Treatment continues every 3 weeks for 4 courses.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
  Arms: Arm II (surgery, chemotherapy)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Arm II (surgery, chemotherapy)
Procedure: therapeutic conventional surgery — Undergo surgery

SUMMARY:
Randomized phase III trial to compare the effectiveness of surgery with or without combination chemotherapy in treating patients who have stage I non-small cell lung cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether surgery is more effective with or without chemotherapy for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if adjuvant chemotherapy can favorably alter the prognosis of the subgroup of resected stage I patients who, following complete surgical resection of their disease, are defined as "high risk" based on the presence of a T2N0 tumor (according to the criteria of the International Staging System for lung cancer).

SECONDARY OBJECTIVES:

I To compare failure-free survival of patients with T2N0 stage I NSCLC who have and have not been treated with adjuvant chemotherapy.

II. To determine the toxicities associated with adjuvant chemotherapy. III. To describe the pattern of disease recurrence.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor histology (squamous cell vs nonsquamous cell), degree of differentiation (poorly differentiated vs other), and mediastinal node sampling at surgery (yes vs no). Within 4-8 weeks after surgery, patients are randomized to 1 of 2 treatment arms.

Arm I:Patients receive no further therapy.

Arm II: Patients receive adjuvant therapy comprising paclitaxel IV over 3 hours followed by carboplatin IV over 1-2 hours on day 1. Treatment continues every 3 weeks for 4 courses.

Patients are followed every 4 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented non-small cell carcinoma
* Completely resected T2N0M0 Stage I NSCLC as defined by the International Staging System
* Surgery shall consist of a lobectomy or pneumonectomy with resection of associated N1 lymph nodes (either by thoracotomy or thoracoscopy)
* Patients must be randomized within 4 to 8 weeks from the date of complete surgical resection
* No prior chemotherapy or radiation for non-small cell lung cancer
* Performance status of 0 or 1
* Women must be non-pregnant and non-lactating; patients of childbearing potential must agree to use an effective form of contraception while on study
* Patients must have no history of previous or concomitant malignancy, other than curatively treated carcinoma in situ of the cervix, or basal cell or squamous cell carcinoma of the skin, or surgically treated in situ carcinoma of the breast, or other cancer for which the patient has bee disease free for five years
* Granulocytes >= 1,800/ul
* Platelets >= 100,000/ul
* Bilirubin < 1.5 mg/dl
* SGOT (AST) < 2.0 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 1996-10; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 2.4 years
  OS curves will be calculated using the Kaplan-Meier life-table method. Comparison of the survival curve for the two treatment regimens will be performed using the log-rank test for censored data.
Failure-free survival | Time between randomization and disease relapse or death, assessed up to 2.4 years
  Failure-free survival curves will be calculated using the Kaplan-Meier life-table method.

SECONDARY OUTCOMES:
Toxicity as assessed by Common Toxicity Criteria version 2.0 | Up to 1 year after completion of treatment
Pattern of disease recurrence. | Up to 2 years
  The frequency of local and distant relapse and the incidence of a second primary lung cancer will be tabulated by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Strauss, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States